CLINICAL TRIAL: NCT02490215
Title: Epidemiology of Acute Respiratory Distress Syndrome in Chinese ICUs
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MICU2015_1
Record Dates: First submitted 2015-05-18; First posted 2015-07-03 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2015-01

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ARDS, non-ARDS: patients with ARDS and patients without ARDS

SUMMARY:
The acute respiratory distress syndrome(ARDS)has a high morbidity and mortality in patients admitted to intensive care units(ICUs). It represents a significant public health issue. No large nationwide, multicenters study of ARDS has been conducted in China. The purposes of this study are to analyse: 1)the incidence and outcomes of ARDS in ICU; 2) factors associated the mortality ; and 3) risk factors for development of ARDS .

DETAILED DESCRIPTION:
All patients admitted to the participating ICUs during a 6-month period(from January 1, 2015 to July 1,2015 ) will be screened at ICU admission and daily for the occurrence of ARDS ( AECC criteria) for a maximum of 28 days after ICU admission.

Data collection:

1. For all patients, Demographic characteristics, admission category, the patient source intervention during ICU , APACHEII , SOFA score and discharge information will be collected
2. For patients with ARDS, data about ABG , parameters of MV, hemodynamic on day0 to day7 and last day of MV will be collected.
3. For patients without ARDS at ICU admission, data about risk factor for ARDS ,such as LIPS score, parameters of MV , and fluid balance on ICU day0 to day7 will be collected.

ELIGIBILITY:
Inclusion Criteria:

all patients age >18 yrs admitted to 24 participating ICUs

Exclusion Criteria:

No patients should be excluded (regardless of age, underlying disease, life expectancy, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the participating ICUs during a 6-month period(from January 1, 2015 to July 1,2015 )
Sampling Method: Non-Probability Sample
Enrollment: 2530 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
incidence of acute respiratory distress syndrome (ARDS) | from ICU admission to 28-day of ICU stay
  incidence of ARDS = the number of patients developing ARDS during ICU / the total number of patients admitted to ICU

SECONDARY OUTCOMES:
ICU mortality of patients with ARDS | followed up to 3 months after inclusion or to ICU discharge, whichever occurred first
hospital mortality of patients with ARDS | followed up to 3 months after inclusion or to hospital discharge, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, Principal Investigator — MICU of Peking Union Medical College Hospital
Locations (26):
- China (26):
  - MICU, Peking union medical college hospital, Beijing, Beijing Municipality
  - Beijing Hospital of ministry of Health, Beijing, Beijing Municipality
  - Department of Critical Care Medicine, Fuxing Hospital, Capital Medical University, Beijing, Beijing Municipality
  - General ICU, Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijng, Beijing Municipality
  - Department of Emergency and Intensive Care Medicine, The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Department of CriticalCare Medicine, Guangdong General Hospital, Guangzhou, Guangdong
  - Department of Critical Care Medicine, Hainan Provincial People's Hospital, Haikou, Hainan
  - Department of Critical Care Medicine, Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - Department of Critical Care Medicine, The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - ICU, The First Affiliated Hospital, Zhengzhou University, Zhengzhou, Henan
  - Department of Critical Care Medicine, Tongji Hospital of Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Department of Critical Care Medicine, Xiangya Hospital, Central South University, Changsha, Hunan
  - Department of Critical Care Medicine, The Affiliated Hopsital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Department of Critical Care Medicine, The Second Hospital of Jilin University, Changchun, Jilin
  - Department of Critical Care Medicine, The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Department of Critical Care Medicine, Qilu Hospital of Shandong University, Jinan, Shandong
  - Emergency ICU, Ruijin Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Surgical Intensive Care Unit, Xijing Hospital, XiAn, Shanxi
  - Department of Critical Care Medicine, West China Hospital, Sichuan University, Chengdu, Sichuan
  - Department of Critical Care Medicine, First Affiliated Hospital, Xinjiang Medical University, Ürümqi, Xinjiang
  - Department of Emergency Medicine and Medical ICU, The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Department of Critical Care Medicine, Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang